CLINICAL TRIAL: NCT05614791
Title: Evaluation of Pediatric Measles Cases in 2019: Single-Center Experience
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, mahmut caner us, M.D, Marmara University
Other Study IDs: 2019.10.2.02.075
Record Dates: First submitted 2022-11-06; First posted 2022-11-14 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2022-11

CONDITIONS: Measles
Keywords: Measles; Vaccine; Children; Vitamin A
MeSH Terms: conditions — Measles

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Measles, can be prevented and eliminated by vaccination, is a highly contagious viral disease that can lead to serious complications, disability, and death. As a result of the World Health Organization (WHO) and United Nations International Children's Emergency Fund (UNICEF) strategic plans, the annual global incidence of measles decreased by 75% over the period 2000-2015, and the estimated global mortality rate fell by 73%. For the current 2019 period, the European and the Eastern Mediterranean Region has recorded respectively more than two-fold and 1.5-fold increase in reported measles cases. As it is known, no specific antiviral treatment exists for the measles virus therefore, vaccination is still the most effective method of preventing disease.

The aim of this study was to evaluate the measles cases in districts where the refugees live quite intensely.

DETAILED DESCRIPTION:
Measles, can be prevented and eliminated by vaccination, is a highly contagious viral disease that can lead to serious complications, disability, and death. As a result of the World Health Organization (WHO) and United Nations International Children's Emergency Fund (UNICEF) strategic plans, the annual global incidence of measles decreased by 75% over the period 2000-2015, and the estimated global mortality rate fell by 73%. For the current 2019 period, the European and the Eastern Mediterranean Region has recorded respectively more than two-fold and 1.5-fold increase in reported measles cases. As it is known, no specific antiviral treatment exists for the measles virus therefore, vaccination is still the most effective method of preventing disease.

The aim of this study was to evaluate the measles cases in districts where the refugees live quite intensely.

This retrospective study was consecutively enrolled children who were considered as suspicious measles case according to with clinical features and attended in Esenler Gynecology and Pediatrics Hospital Pediatric Clinic between 01 January-30 June 2019.

ELIGIBILITY:
Inclusion Criteria:

* The suspicious case of measles
* Measles/Rubella Case Notification and Laboratory request and result form and Measles/ Rubella Case Study form must be filled
* Accept the informed consent form
* Positive Measles Ig M and Measles Ig G laboratory test

Exclusion Criteria:

* Rejected the informed consent form

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Measles case according to with clinical features and attended Pediatric Clinic between 01 January-30 June 2019
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of measles vaccination status on symptom duration | baseline
  compare the groups symptom durations (day) who fully, partly or not vaccinated
Evaluate the effect of vitamin A treatment on symptom duration | in the first month after the first symptom observed
  compare the groups symptom durations (day) who get or not get vitamin A treatment

SECONDARY OUTCOMES:
Evaluate the effect of measles vaccination status on leucocyte count | baseline
  compare the groups leucocyte count who fully, partly or not vaccinated
Evaluate the effect of vitamin A treatment on leucocyte count | baseline
  compare the groups leucocyte count who get or not get vitamin A treatment

OTHER OUTCOMES:
Evaluate the effect of measles vaccination status on cost of measles cases | in the first month after the first symptom observed
  compare the groups costs (Turkish Lira) who fully, partly or not vaccinated
Evaluate the effect of vitamin A treatment on cost of measles cases | in the first month after the first symptom observed
  compare the groups costs (Turkish Lira) who get or not get vitamin A treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Caner US, MD, Principal Investigator — haseki Education and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Esenler Maternity and Child Health Hospital, Istanbul, Esenler
  - Haseki Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided
Availability of data and material: When needed, all data can be shared with the consent of the participants.

REFERENCES:
- [Background] Lord H, Kok J, Fletcher S, Alexander K. Is it or is it not? Lessons learned from a case of suspected vaccine strain measles. Aust N Z J Public Health. 2020 Apr;44(2):160-162. doi: 10.1111/1753-6405.12969. Epub 2020 Mar 19. PMID 32190947
- [Background] Lo Vecchio A, Krzysztofiak A, Montagnani C, Valentini P, Rossi N, Garazzino S, Raffaldi I, Di Gangi M, Esposito S, Vecchi B, Melzi ML, Lanari M, Zavarise G, Bosis S, Valenzise M, Cazzato S, Sacco M, Govoni MR, Mozzo E, Cambriglia MD, Bruzzese E, Di Camillo C, Pata D, Graziosi A, Sala D, Magurano F, Villani A, Guarino A, Galli L; SITIP Measles Study Group. Complications and risk factors for severe outcome in children with measles. Arch Dis Child. 2020 Sep;105(9):896-899. doi: 10.1136/archdischild-2018-315290. Epub 2019 Jan 12. PMID 30636224
- [Background] Filia A, Bella A, Del Manso M, Baggieri M, Magurano F, Rota MC. Ongoing outbreak with well over 4,000 measles cases in Italy from January to end August 2017 - what is making elimination so difficult? Euro Surveill. 2017 Sep 14;22(37):30614. doi: 10.2807/1560-7917.ES.2017.22.37.30614. PMID 28933342